CLINICAL TRIAL: NCT00429611
Title: A Multicentre Prospective Randomised Study Comparing the Efficacy of High Versus Low Biphasic Energy Defibrillation in Patients With Cardiac Arrest
Brief Title: High Low Biphasic Energy Defibrillation (HiLoBED)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Medtronic (Industry); National Heart Centre Singapore (Other); Tan Tock Seng Hospital (Other); Changi General Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Prof. V. Anantharaman, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SQCA02
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Ventricular Fibrillation
Keywords: biphasic defibrillation; inhospital; post-resuscitation myocardial function; defibrillation efficacy; high energy versus low energy; cardiac arrest patients
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cardiac defibrillation at high energy vs low energy levels — Defibrillation with progressive high-energy biphasic shocks at 200J, 300J and 360J or low-energy biphasic shocks at 150J, 150J and 150J.

SUMMARY:
This inhospital study aims to compare the efficacy of high-versus low-energy biphasic shocks in order to determine the optimal level for defibrillation. Time is the essence when attending to a VF patient. Hence, it is important to determine the optimal amount of defibrillation energy that should be delivered at first shock, thereby increasing the patient's chances of survival. In addition, this study provides an opportunity to evaluate the impact on myocardial integrity/function of different levels of defibrillation energy in an inhospital clinical environment.

DETAILED DESCRIPTION:
This is a prospective, randomised study to be conducted in the Emergency Medicine Departments and Cardiology Departments of four major hospitals, viz. Singapore General Hospital, National University Hospital, Changi General Hospital and Tan Tock Seng Hospital. The four hospitals were selected as they generally handle the most patients experiencing ventricular fibrillation (VF) and pulseless ventricular tachycardia (VT) in the inhospital setting in this country. The study will include patients with cardiac arrest, who have a shockable rhythm (VF and pulseless VT) and aged 21 years and above. Patients who have received defibrillation pre-hospital will also be included if they are still in VF at time of arrival at the hospital.

Patients will be administered one of the following:

* Defibrillation with progressive high-energy biphasic shocks using the Medtronic Physio-Control LifePak 12 at 200J, 300J and 360J. If still unsuccessful, further shocks at 360J plus anti-arrhythmics as per American Heart Association (AHA) and Singapore National Resuscitation Council (NRC) guidelines for mega VF will be applied.
* Defibrillation with low-energy biphasic shocks using the Medtronic Physio- Control LifePak 12 at 150J, 150J and 150J. If still unsuccessful, shocks will be continued at the higher energy range (as above) plus the use of anti- arrhythmics as per the AHA and NRC guidelines for mega VF.

Results will be analysed to obtain first/subsequent shock defibrillation efficacy and post-shock myocardial function/dysfunction. This randomised study is the first of its kind to explore the efficacy of different biphasic energy levels and their impact on myocardial integrity/function in an inhospital clinical setting. After completion, the study will be expected to produce at least Level 2 results, which would be useful to international resuscitation committees in determining future guidelines and recommendations for defirillation in cardiac arrest victims.

At the conclusion of the study, the results will be analysed and published as soon as possible. This will be the responsibility of the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* patients with cardiac arrest, who have a shockable rhythm (ventricular fibrillation and pulseless ventricular tachycardia)
* aged > or equal to 21 years

Exclusion Criteria:

* aged below 21 years (young patients whose ages cannot be determined accurately will not be included)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2004-11; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Return of Spontaneous Circulation (ROSC) | First shock ROSC

SECONDARY OUTCOMES:
Survival at 24 hours, 7 and 30 days | 24 hours after defibrillation, seven days and 30 days after admission
Myocardial damage/dysfunction as indicated by ST segment elevation/depression (mm) at 1 minute, 10 minutes and 24 hours, highest CKMB level and LVEF by echocardiography. | within 24 hours of defibrillation

CONTACTS AND LOCATIONS:
Overall Officials: V Anantharaman, MBBS, Principal Investigator — Singapore General Hospital
Locations (7):
- Singapore (7):
  - Accident and Emergency Department, Changi General Hospital, Singapore
  - Department of Cardiology, Tan Tock Seng Hospital, Singapore
  - Department of Emergency Medicine, Singapore General Hospital, Singapore
  - Division of Cardiology, Changi General Hospital, Singapore
  - Division of Cardiology, National Heart Centre, Singapore
  - Emergency Medicine Department, National University Hospital, Singapore
  - Emergency Medicine Department, Tan Tock Seng Hospital, Singapore